CLINICAL TRIAL: NCT00232739
Title: A Multicenter, Non-Randomized Study of the 2.25mm Sirolimus-Eluting BX VELOCITYTM Balloon-Expandable Stent in the Treatment of Patients With de Novo Native Coronary Artery Lesions
Brief Title: Study of the 2.25mm Sirolimus-Eluting Stent in the Treatment of Patients With Coronary Artery Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Sriram Iyer, MD, Lenox Hill Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03-6320
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2010-02-08 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2010-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: CYPHER Sirolimus-eluting Coronary Stent

INTERVENTIONS:
Device: CYPHER Sirolimus-eluting Coronary Stent — 2.25 Cypher Sirolimus-eluting Coronary Stent

SUMMARY:
The main objective of this study is to assess the safety and effectiveness of the sirolimus-eluting Bx VELOCITYTM stent in reducing in-lesion restenosis in patients with de novo native coronary artery lesions.

DETAILED DESCRIPTION:
This is a multicenter (approximately 10 - 14 sites), prospective, non-randomized study. The study is designed to evaluate the safety and effectiveness of the sirolimus-eluting Bx VELOCITYTM stent in patients with de novo native coronary artery lesions. A total of 100 patients will be entered in the study. Patients who meet the eligibility criteria will be enrolled into the study. Patients will be followed at 30 days, 6, 9, and 12 months, and at 2, 3, 4 and 5 years post-procedure, with all patients undergoing repeat angiography at 6 months. Approximately 50 patients will be required to have an intravascular ultrasound (IVUS) procedure at baseline and at the 6-month angiographic follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant female patients minimum 18 years of age
2. Diagnosis of angina pectoris as defined by Canadian Cardiovascular Society Classification (CCS I, II, III, IV) OR unstable angina pectoris (Braunwald Classification B&C, I-II) OR patients with documented silent ischemia;
3. Target lesion is 20mm in length (visual estimate);
4. Target lesion stenosis is >50% and <100% (visual estimate);

Exclusion Criteria:

1. Patient has experienced a Q-wave or non-Q-wave myocardial infarction with documented total CK >2 times normal within the preceding 24 hours and the CK and CK-MB enzymes remains above normal at the time of treatment;
2. Has unstable angina classified as Braunwald III B or C, or is having a peri infarction;
3. Documented Left ventricular ejection fraction 25%;
4. Impaired renal function (creatinine > 3.0 mg/dl) at the time of treatment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2003-09; Primary Completion 2004-11 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Iyer, MD, Principal Investigator — Lenox Hill Hospital
Locations (1):
- Lenox Hill Hospital, New York, New York, United States

REFERENCES:
- [Background] Moses JW, Nikolsky E, Mehran R, Cambier PA, Bachinsky WB, Leya F, Kuntz RE, Popma JJ, Schleckser P, Wang H, Cohen SA, Leon MB; SIRIUS 2.25 Investigators. Safety and efficacy of the 2.25-mm sirolimus-eluting Bx Velocity stent in the treatment of patients with de novo native coronary artery lesions: the SIRIUS 2.25 trial. Am J Cardiol. 2006 Dec 1;98(11):1455-60. doi: 10.1016/j.amjcard.2006.06.047. Epub 2006 Oct 13. PMID 17126649

RESULTS

PARTICIPANT FLOW:
Groups:
- 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent: The 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-expandable stent in patients with de novo native coronary artery lesions
Period: Overall Study
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Started | 100
Completed | 91
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 63.4 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 64
Region of Enrollment [Number; unit: participants]
  United States | 100
Diabetes Mellitus [Number; unit: participants]
  Diabetes Mellitus | 40
  Without Diabetes Mellitus | 60 [30.3 to 50.3]
History of Myocardial Infarction (MI) [Number; unit: participants]
  History of MI | 33 [25.5 to 45.6]
  Without History of MI | 61
  N/A | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced In-lesion Restenosis as Measured by Quantitative Coronary Angiography (QCA) at 6 Months Post-procedure
Description: In-lesion restenosis was defined as over 50 percent diameter stenosis either within the stented segment or within 5 mm proximal or distal to the stent edges at a qualifying follow-up angiogram.
Time Frame: From post-procedure to 6 months
Population: The number of participants with six months follow up and non-missing six months binary angiographic restenosis (BAR) results.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 77
Percentage of participants | 16.9 [9.3 to 27.1]
Statistical Analysis 1: Comparison: 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent; Historical control groups consist of propensity-scored matched cohorts (100 patients each, based on Reference Vessel Diameter, lesion length, diabetes, left anterior artery diseased vessel, and gender) of plain old balloon angioplasty (POBA), first generation (Palmaz-Schatz) bare metal stent (BMS1), and BX VELOCITY bare metal stent (BMS2). Study showed the risk of 6-month in-lesion binary angiographic restenosis (BAR) was much lower for the 2.25 Sirolimus stent compared with POBA, BMS1 or BMS2; Test type: Superiority or Other; Bayesian regression model — The primary analysis of comparing Sirolimus stent with POBA using Bayesian regression model yields that Sirolimus is superior to POBA in reducing the BAR risk; Multi-level Bayesian regression model was used in the secondary analysis; Primary analysis posterior probability = 0.9926 — Secondary analysis for comparing Sirolimus stent with BMS1 and BMS2 signified that Sirolimus stent is superior to POBA, BMS1 and BMS2 in reducing the BAR risk

2. Secondary Outcome: Cumulative Percentages of Participants Who Experienced Any Major Adverse Cardiac Events up to Each Scheduled Follow-up
Description: The percentages are cumulative up to each of the scheduled post-procedure follow-up: 30 days, 6, 9, and 12 months, and 2, 3, 4 and 5 years. Major Adverse Cardiac Events (MACE) consists of death, Myocardial Infarction (Q-wave and Non Q-wave), emergent Coronary Artery Bypass Graft (CABG) or Target Lesion Revascularization (TLR).
Time Frame: From post-procedure to 4 years
Population: The number of participants who had four years post-procedure follow up or who had at least one event prior to the end of follow-up.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 96
Percentage of participants
  6 Months Post-Procedure | 8.0 [2.7 to 13.3]
  9 Months Post-Procedure | 9.0 [3.3 to 14.7]
  12 Months Post-Procedure | 11.0 [4.9 to 17.1]
  2 Years Post-Procedure | 17.0 [9.6 to 24.4]
  3 Years Post-Procedure | 21.0 [13.0 to 29.0]
  4 Years Post-Procedure | 27.4 [18.2 to 36.6]

3. Secondary Outcome: Percentage of Participants Who Experienced Any Angiographic In-stent Binary Restenosis up to 6 Months Post-procedure.
Description: In-stent restenosis was defined as greater than or equal 50 percent diameter stenosis within the stented segment at a qualifying follow-up angiogram.
Time Frame: From post-procedure to 6 months
Population: The number of participants with six months follow up and non-missing six months binary angiographic restenosis results.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 77
Percentage of participants | 11.7 [5.5 to 21.0]

4. Secondary Outcome: Average In-stent and In-lesion Minimum Lesion Diameters (MLD) at 6 Months Post-procedure.
Time Frame: From post-procedure to 6 months
Population: The number of participants with six months follow up and non-missing six months binary angiographic restenosis results.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 77
mm
  Average In-stent MLD | 1.64 (0.52)
  Average In-lesion MLD | 1.35 (0.45)

5. Secondary Outcome: Cumulative Percentages of Participants Who Experienced Any Target Lesion Revascularization (TLR) up to 6 and 9 Months Post-procedure.
Description: TLR was defined as any "clinically-driven" repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel.
Time Frame: From post-procedure to 6 months and 9 months
Population: The number of participants who had sufficient follow-up or who had an event prior to the end of follow-up.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 95
Percentage of participants
  6 Months Post-Procedure | 5.1 [0.8 to 9.4]
  9 Months Post-Procedure | 6.1 [1.2 to 11.0]

6. Secondary Outcome: Cumulative Percentages of Participants Who Experienced Any Target Vessel Revascularization (TVR) up to 6 and 9 Months Post-procedure.
Description: TVR was defined as any clinically driven repeat percutaneous intervention of the target vessel or bypass surgery of the target vessel. Clinically-driven revascularizations were those in which the patient has a positive functional study, ischemic ECG changes at rest in a distribution consistent with the target vessel, or ischemic symptoms, and an in-lesion diameter stenosis being greater than or equal to 50 percent measured by QCA.
Time Frame: From post-procedure to 6 months and 9 months follow-up
Population: The number of participants who had sufficient 9 months post-procedure follow-up or had the event prior to 9 months.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 95
Percentage of participants
  6 Months Post-Procedure | 8.1 [2.8 to 13.4]
  9 Months Post-Procedure | 10.1 [4.2 to 16.0]

7. Secondary Outcome: Cumulative Percentages of Participants Who Experienced Any Target Vessel Failure (TVF) up to 6 and 9 Months Post-procedure
Description: TVF was defined as any Target vessel revascularization, Q wave or non-Q wave MI, or cardiac death that could not be clearly attributed to a vessel other than the target vessel.
Time Frame: From post-procedure to 6 months and 9 months follow-up
Population: The number of participants who had sufficient follow-up or who had an event prior to the end of follow-up.
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 96
Percentage of participants
  6 Months Post-Procedure | 11.0 [4.9 to 17.1]
  9 Months Post-Procedure | 13.0 [6.3 to 19.7]

8. Secondary Outcome: Average Lumen Volume (mm3) at Post-procedure
Time Frame: At Post-procedure
Population: The number of participants who had lumen volume data at post-procedure
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 11
mm3 | 73.34 (38.32)

9. Secondary Outcome: Average Stent Obstruction Volume at Post-procedure
Description: Stent obstruction Volume equals 100 * [1-(lumen volume/baseline stent volume)]; usually this is equal to zero at baseline, since the stent is freshly implanted and no obstruction is expected
Time Frame: At post-procedure
Population: Number of participants who had Stent Obstruction Volume data at post-procedure
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 11
mm3 | 0.0 (0.0)

10. Secondary Outcome: Average Lumen Volume (mm3) at 6 Months Post-procedure
Time Frame: From post-procedure to 6 months
Population: The number of participants who had Lumen Volume data at 6 months post-procedure
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 8
mm3 | 70.25 (25.61)

11. Secondary Outcome: Average Stent Obstruction Volume at 6 Months Post-procedure
Time Frame: From post-procedure to 6 months
Population: The number of participants with Stent Obstruction Volume data at 6 months post-procedure
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 8
mm3 | 3.05 (2.42)

12. Secondary Outcome: Percentage of Participants Who Achieved Lesion Success at Post-procedure
Description: Lesion success defined as the attainment of <50 percent residual stenosis (by QCA) using any percutaneous method
Time Frame: At post-procedure
Population: Number of Participants without missing lesion success data
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 99
Percentage of participants | 98.0 [92.9 to 99.8]

13. Secondary Outcome: Percentage of Participants Who Achieved Device Success at Post-procedure
Description: Device success was defined as achievement of a final residual diameter stenosis of less than 50 percent as measured by QCA, using the assigned device only. If QCA is not available, the visual estimate of diameter stenosis is used
Time Frame: At post-procedure
Population: All participants
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 100
Percentage of participants | 96.0 [90.1 to 98.9]

14. Secondary Outcome: Percentage of Participants Who Achieved Procedure Success Before Hospital Discharge
Description: Procedure success defined as achievement of a final diameter stenosis of less than 50 percent (by QCA) using any percutaneous method, without the occurrence of death, MI, or repeat revascularization of the target lesion during the hospital stay
Time Frame: From post-procedure to hospital discharge
Population: Number of participants without missing procedure success data
Measure: Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Number analyzed (Participants) | 99
Percentage of participants | 97.0 [91.4 to 99.4]

ADVERSE EVENTS:
Time Frame: From post-procedure to 1440 days follow up
Arm/Group | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent
Serious Adverse Events (participants affected / at risk) | 5/91
Other Adverse Events (participants affected / at risk) | 39/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent (N=91)
Death (Vascular disorders) | 5 (5) — Total number of participants who died from post-procedure to 1440 days follow up.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 2.25mm Sirolimus-eluting Bx VELOCITY™ Balloon-exp Stent (N=96)
Myocardial Infarction (Q wave or Non-Q wave) (Vascular disorders) | 14/94 (14) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Target Lesion Revascularization (Vascular disorders) | 14/95 (14) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Target Vessel Revascularization not involving Target Lesion (Vascular disorders) | 8/92 (8) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Target Vessel Revascularization (All) (Vascular disorders) | 20/95 (20) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Acute/Subacute Stent Thrombosis to 30 Days (Vascular disorders) | 1/92 (1) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Late Stent Thrombosis (31-1440 Days) (Vascular disorders) | 4/91 (4) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Subacute Closure (Vascular disorders) | 1/92 (1) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Cerebrovascular Accident (CVA) (Vascular disorders) | 4/92 (4) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Hemorrhagic Vascular Complications (Vascular disorders) | 6/92 (6) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up
Target Vessel Failure (Vascular disorders) | 26 (26) — The number at risk is defined as the number of participants who had sufficient 4 years post-procedure follow-up or who had at least one event prior to the end of follow-up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days